CLINICAL TRIAL: NCT06165471
Title: The Effectiveness of a Mobile Application for Teaching Clinical Nursing Skill at a Higher Education Institution in Chenzhou, China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, LI AFANG, Doctor of Philosophy student, Nursing Education, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: USM/JEPeM/KK/23020172
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Nursing Education
Keywords: Pretest-post test and intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended learning group (Experimental): The Intervention group will adopt the mode of online and offline blended learning based on the Chaoxing mobile application (Chaoxing app). The researchers will create surgical nursing practice courses on the Chaoxing app, and the experimental group will be subjected to 2 months of online and offline blended teaching intervention using the Chaoxing app.
  Interventions: Behavioral: Online and offline blended teaching
- Traditional teaching group (Active Comparator): The control group will adopt the traditional face-to-face teaching method for the surgical nursing practice course. The teacher will demonstrate the process, and the students will practice. The teacher demonstrates each step, and the students practice each step.
  Interventions: Behavioral: Traditional teaching

INTERVENTIONS:
Behavioral: Online and offline blended teaching — The Chaoxing app is an interventional tool, a professional mobile learning platform for smartphones, tablet computers, and other mobile terminals. They will learn the online course on the Chaoxing app and carry out offline classroom learning. The online courses focus on teaching design to make teaching PowerPoint, teaching videos, micro-lessons, homework library, and so on.
  Arms: Blended learning group
Behavioral: Traditional teaching — The researchers will implement the traditional teaching intervention of a surgical nursing practice course to the control group, and the teacher will demonstrate the operation procedure to the students face to face offline, and the students will practice. The whole intervention time is two months.
  Arms: Traditional teaching group

SUMMARY:
The general objective of this study is to validate a mobile application as a pedagogical tool compared to in-person nursing educational instruction for teaching clinical nursing skills and evaluate the effectiveness of clinical nursing skills for nursing students.

The study design is a basic experimental study design, randomized control trial (RCT) design; the dependent variables measured in this study are skills, self-directed learning ability, online academic emotion, and satisfaction by using pre- and posttests; two groups are participating in this study; experimental and control group. The control group treatment is traditional face-to-face teaching, and the experimental group intervention is online and offline blended learning based on the Chaoxing app. The study process includes four steps：

1. To develop surgical nursing practical online courses using Chaoxing mobile app.
2. Perform the pre-test (basic sociological information, self-directed learning ability surveys ).
3. Nursing clinical practice skills education intervention.
4. Perform a posttest (assess practical skills, self-directed learning ability, online academic emotion, and satisfaction).

DETAILED DESCRIPTION:
Study title:

The Effectiveness of A Mobile Application for Teaching Clinical Nursing Skill at A Higher Education Institution in Chenzhou, China

General objective:

The general objective of this study is to validate a mobile application as a pedagogical tool compared to in-person nursing educational instruction for teaching clinical nursing skills and evaluate the effectiveness of clinical nursing skills for nursing students.

The study design is a basic experimental study design, randomized control trial (RCT) design; the dependent variables measured in this study are skills, self-directed learning ability, online academic emotion, and satisfaction by using pre- and posttests; two groups are participating in this study; experimental and control group. The control group treatment is traditional face-to-face teaching, and the experimental group intervention is online and offline blended learning based on the Chaoxing app. The study process includes four steps：

1. To develop surgical nursing practical online courses using the Chaoxing mobile app.
2. Perform the pre-test (basic sociological information, self-directed learning ability surveys ).
3. Nursing clinical practice skills education intervention.
4. Perform a posttest (assess practical skills, self-directed learning ability, online academic emotion, and satisfaction).

Study Location:

This study will be conducted at Xiangnan University in Chenchou city Hunan province in China, Chenzhou city is in the southeast of China.

Study Design:

The study design was a prospective, single-blind experimental design, randomized control trial (RCT) design.

Study population & Setting The sample will consist of third-year undergraduate nursing students at a university in Chenzhou, southeast China. They are between 19 and 22 years old. In the early stage, students have completed one year of basic medical courses and mastered the relevant knowledge of human anatomy, physiology, and pathology. Students are active in thinking, have intense curiosity, and have a certain ability to understand and self-learning. However, students are exposed to clinical practice skills for the first time and have little exposure to clinical practice in the early stage, resulting in poor comprehensive analysis ability and unfamiliar skills operation.

Sample size calculation:

The sample size estimate was calculated based on the primary measure of self-learning ability. Sample size calculation is performed by using G*POWER software (version 3.1.9.4) and consists of the following steps: (1) Select the test family (t-test ), (2) Select the statistical test (Means: Difference between two independent means (two groups)), (3) Select the Type of power analysis (A priori: Compute required sample size - given α, power, and effect size), (4) Select tails (two), α err prob (0.05), Power (1-β err prob) (0.95), Allocation ratio N2/N1 is one (each group = n) n= the estimated sample size. Effect Size (ES) = 0.55, automatically calculated by G*Power software, depending on the sample size of the previous studies (Luo Qiaoling, 2020) ,(Zhang Y H,2015),(Li X M, 2021), the effect size is calculated by selecting these similar studies fitted to the researchers' study, the reasonable sample size which is (n=166) will be taken as the minimum sample size for this study, and the minimum sample size for each group will be 83 participants.

Sampling method:

Cluster random sampling was used after obtaining ethical approval and permission to conduct the study from the Ethics Committee of Xiangnan University, China (Ethics Registration No. 2022YXLL030) and the Jawatankuasa Etika Penyelidikan Manusia, Universiti Sains Malaysia (JEPeM-USM), the study protocol code USM/JEPeM/KK/23020172. The cluster sampling method of the participants was used to select all the undergraduate students in 2021 from the School of Nursing of Xiangnan University, Chenzhou, China. Computer-generated randomization (Random Allocation Software, version 1.0) was applied in blocks to allocate the classes by distributing them into two arms: one is the control group, and the other is the experimental group.

Study process steps:

(i) In the Pre-Test, the estimated time to fill will be 15 minutes maximum; it consists of 2 sections. The first section includes the consent form and ten questions about demographical data; the second section includes a self-directed learning ability assessment and consists of 20 MCQ questions. The pre-test will be filled out by both the control and interventional groups.

(ii) The intervention, volunteer participation, takes about two months for both the control and interventional groups. The control group will adopt the traditional face-to-face teaching mode, and the interventional group will adopt the mode of online and offline blended learning based on the Chaoxing app.

(iii) In the post-test, the interventions are finished, and an examination evaluation will be immediately given to both group's participants, including online academic emotional, self-directed learning ability, and class satisfaction assessment with a total of 55 MCQ questions, which will be 30 minutes maximum.

Ethical Considerations：

1. Permission to conduct the study Regarding ethical considerations, approval for the study was obtained from the Jawatankuasa Etika Penyelidikan Manusia, Universiti Sains Malaysia (JEPeM-USM), the study protocol code USM/JEPeM/KK/23020172; Moreover, ethical approvals to conduct the study was obtained from the Ethics Committee of Xiangnan University, China (Ethics Registration No. 2022YXLL030).
2. Subject vulnerability: Participants will be informed of their right to participate voluntarily and to withdraw from the study at any time without being penalized or losing the benefits to which they would otherwise be entitled. Informed consent was signed after all procedures were explained to each participant, and they agreed to participate in the study. For participants who need clarification on the study, the researchers will detail the instructions so that they fully understand and then agree to participate. During this study, the researcher is not a teacher as she is on study leave and not doing any teaching work. She is a researcher who will conduct the study and recruit the students. All teaching processes and materials will be handled by the teaching team. The researcher will not affect the student's evaluation during the study period.
3. Privacy and confidentiality: All personal data, including consent forms and questionnaire data obtained from study participants, will be kept strictly confidential and used only for academic and research purposes. In addition, the subject's name will not appear on any documents to maintain anonymity.
4. Conflict of interest: The principal investigator is the teacher in the faculty where data collection takes place; there are no conflicts of interest in the study, nor was there anything that might affect or prejudice the professional judgment in the study.
5. Community sensitivities and benefits: This study does not have any relation with sensitivity to the community because this study only involves a student and the impact of the technology used for their education. If the student uses the technology for nursing education, the benefit will go to the students directly. At the end of the study, the control group could also use the online course on the Chaoxing app if proven effective.
6. Incentive, compensation &/or reimbursement: Participants in this study do not incur any fees. The study will not offer any monetary or other rewards in response to participation.
7. The risks in this study: The study was free from any potential hazards or adverse effects on participants; no dedicated product will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* i) Full-time undergraduate nursing students in grades 3 who understand Chinase language.
* ii) Owning at least one smartphone, tablet or portable laptop.

Exclusion Criteria:

* i) Repeat students.
* ii) Sick (matter) leave, Suspension of schooling.
* iii) Can not fully participate in or cooperate with.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
The effects of surgical nursing practical online courses using Chaoxing app on the skills score | Hence the interventions finished, and an examination evaluation will be immediately given to the both groups participants.
  Skill test will be given after both groups students have completed the course. The same academic grading scale will be used for both groups that formulated with the approval of the Teaching and Research Section. Exam scores will only be used for this study, It will not impact the score or grading of the students and do not serve as a final grade of the student.
Self-directed learning ability | Hence the interventions finished, and an examination evaluation will be immediately given to the both groups participants.
  The level of Self-directed learning ability will be measured by the Self-Directed Learning Instrument (SDLI) for Nursing Students developed by Cheng S F et al. (Cheng, S. F.,2010) from Taiwan, which is a self-evaluation scale of nursing students' autonomous learning ability. After reliability and validity testing of Chinese version, it popularized and used in Mainland China (Shen, W. Q., 2014). The scale including learning motivation, plan and implement, self management, interpersonal communication, 4 dimensions, a total of 20 items.

SECONDARY OUTCOMES:
Online academic emotional assessment | Hence the interventions finished, and an examination evaluation will be immediately given to the both groups participants.
  The online academic emotion scale was developed by Pekrun(Pekrun R, 2002) et al., introduced by Zhan Yi(Zhan Yi,2016), and later modified by Liu Junling (Liu Junling, 2019)et al., combined with the characteristics of online learning for college students, and finally formed the Online Academic Emotion Scale for College Students. The scale included 3 dimensions, 6 kinds of emotions and 25 items, negative low arousal emotion (8 items), negative high arousal emotion (9 items), positive high arousal emotion (8 items); Likert5-point scoring method was used in the scale, with 1-5 points for "very inconsistent", "inconsistent", "general", "consistent" and "very consistent"; The higher the score of each dimension, the more significant the relevant emotional experience. Validation in Chinese version has been done by Liu Junling, 2019 and the cronbach's α coefficient of the scale was 0.89, and cronbach's a coefficient of each dimension were 0.790-0.897.
Class satisfaction assessment | Hence the interventions finished, and an examination evaluation will be immediately given to the both groups participants.
  The teaching satisfaction evaluation scale was developed by Chinese researcher Fengqin Xu (Xu, 2020) et al.,which, consists of 6 items, Stimulate learning interest and enthusiasm for participation, contribute to knowledge understanding and consolidation of knowledge, help to improve self-learning ability, help Reasonable allocation of time, helpful to the sharing of teaching resources and overall evaluation of the training method. According to the content of this study, the researcher changed the last item overall evaluation of the training method to an overall evaluation of the teaching method. using the Likert 5 scoring method, Very dissatisfied~very satisfied, 0~4 points, total score 0~24 points, total score the higher the score, the more satisfied the respondents are. The cronbach α coefficient of the questionnaire 0.90 and 0.93 for content validity(Xu, 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Afang Li, Principal Investigator — Xiangnan University, China
Locations (1):
- Afang Li, Chenzhou, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Only the participant data related to the study after participate and publication consent without mentioned name, ID, email...and providing the privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after finish and publish the study and will not use in any other study
Access Criteria: Data is kept properly and handled only in the research. In addition, the researchers also emphasized that only research groups can access the relevant data in this research and not use it in the future without consent from the participants; moreover, after finishing the study, the data will archive properly according to the policy.

REFERENCES:
- [Background] Arslan, G. G., Ozden, D., Goktuna, G., & Ayik, C. (2018). A study on the satisfaction of students for the time spent watching video-based learning during their basic nursing skills' training. International Journal of Caring Sciences, 11(1), 427-436.
- [Background] Arguel, A., & Jamet, E. (2009). Using video and static pictures to improve learning of procedural contents. Computers in human behavior, 25(2), 354-359.
- [Background] Chiang, V. C. (2015). Continuous Clinical Assessment (CCA) in Baccalaureate Nursing Education: The Application of Action Research. Journal of Problem-Based Learning, 2(1), 35-47. https://doi.org/10.24313/jpbl.2015.2.1.35.
- [Background] Debande, O., 2004. ICTs and the development of e-learning in Europe: the role of the public and private sectors. European Journal of Education, 39(2) 191-208. https://www.jstor.org/stable/1503883.
- [Background] Duan Zhigang, SUN Hong-yu, LIU Lin. Nursing Education [M].Version5. Beijing: People's Medical Publishing House, 2022.
- [Background] Fox, S., Mckeogh, F., 2003. Can e-learning promote higher-order learning without tutor overload? Open Learning 18(2) 121-134. https://doi.org/10.1080/02680510307410.
- [Background] Goodison, T., 2001. The Implementation of e-learning in higher education in the United Kingdom: The road ahead. Higher Education in Europe, 26(2) 247-262. https://doi.org/10.1080/03797720120082642.
- [Background] Gokcearslan, S. (2017). Perspectives of Students on Acceptance of Tablets and SelfDirected Learning with Technology. Contemporary educational technology, 8(1), 40- 55.
- [Background] Goosen, L., & Van Heerden, D. (2019). Student Support for Information and Communication Technology Modules in Open Distance Environments: Towards SelfDirected Learning. In Student Support Toward Self-Directed Learning in Open and Distributed Environments (pp. 26-58). IGI Global. DOI: 10.4018/978-1-5225-9316-4.ch002.
- [Background] HE Zhijie, Xie Caihong, Chen Ying, Huang Canxia, CAI Qiaowen, Wang Chengling... & Li Fangyi.(2023). Application of online and offline mixed teaching in mechanical ventilation practice teaching of respiratory rehabilitation. Chinese Journal of Rehabilitation Medicine (03),384-387.
- [Background] Huang Yibing. An empirical study on the evaluation of humanistic care ability of nursing college students [D]. Fuzhou: Fujian Medical University,2007.
- [Background] Keller JM. Motivational Design for Learning and Performance: The ARCS Model Approach. New York: Springer; 2010.
- [Background] Li X M, Gao Y, Zheng H P & Zhao J. (2021). The practice of online and offline hybrid assessment of Basic Nursing training based on network platform. Chin J Nursing (17),23-27.Doi:10.16460/ j.isn1008-9969.2021.17.023.
- [Background] Li W. Experimental teaching design and practice of basic Nursing based on the improvement of humanistic care ability of nursing students [D]. Xinxiang: Xinxiang Medical College,2012.
- [Background] Liu Junling, Liu Bin, Zhang Wenlan.(2019). The influence of academic emotion on online collaborative problem solving. China E-Education, (07):82-90.
- [Background] Luo Qiaoling, Li Xiaoping & Wu Jingmei.(2020). The impact of formative assessment based on online learning platform on independent learning of post-secondary nursing students. Journal of Nursing (03),10-13.Doi:10.16460/ j.ssn1008-9969.2020.03.010.
- [Background] MAO Min. Research on piano Teaching Innovation of Young Teachers under the Theory of Independent Learning [D]. Nantong: Nantong University,2015.
- [Background] McKenny, K. (2011). Using an online video to teach nursing skills. Teaching and learning in nursing, 6(4), 172-175. https://doi.org/10.1016/j.teln.2011.04.003
- [Background] Meng Wangtao. Research on the construction and application of the teaching scheme of
- [Background] Pekrun, R., Goetz, T., Titz, W., & Perry, R. P. (2002). Academic emotions in students' self-regulated learning and achievement: A program of qualitative and quantitative research. Educational psychologist, 37(2), 91-105. https://doi.org/10.1207/S15326985EP3702_4
- [Background] Xu Fengqin, Ma Liang, Zhou Guohui, etc. (2020). Newly recruited nurses should Observation on the effect of online and offline pre-employment training. Nursing Journal, (18):21-24
- [Background] Xu Jun, Wan Shuang yan, Liu Xin. (2012). Innovation of clinical basic skills to improve clinical practice ability [J]. Journal of liaoning medical college (social science edition), 10(01):32-34.
- [Background] Zhan Yi. Empirical Research on In-service Teachers' Online Academic Emotions [D]. East China Normal University,2016.
- [Background] Zhang Y H, Zhou Z X, Feng R & Xu H. (2015). Implementation and effect evaluation of flipped classroom for Obstetrics and Gynecology Nursing in higher vocational colleges. Journal of Nursing (06),77-79. Doi:CNKI:SUN:HLXZ.0.2015-06-033.
- [Result] Chen B, Wang Y, Xiao L, Xu C, Shen Y, Qin Q, Li C, Chen F, Leng Y, Yang T, Sun Z. Effects of mobile learning for nursing students in clinical education: A meta-analysis. Nurse Educ Today. 2021 Feb;97:104706. doi: 10.1016/j.nedt.2020.104706. Epub 2020 Dec 5. PMID 33360012
- [Result] Cheng SF, Kuo CL, Lin KC, Lee-Hsieh J. Development and preliminary testing of a self-rating instrument to measure self-directed learning ability of nursing students. Int J Nurs Stud. 2010 Sep;47(9):1152-8. doi: 10.1016/j.ijnurstu.2010.02.002. Epub 2010 Mar 11. PMID 20223455
- [Result] Durmaz Edeer A, Vural F, Turhan Damar H, Yasak K, Damar M. The Effect of Web-Based Preoperative and Postoperative Patient Care Education on Nursing Students: A Randomized Controlled Study. Comput Inform Nurs. 2019 Oct;37(10):541-547. doi: 10.1097/CIN.0000000000000552. PMID 31373901
- [Result] Forman D, Nyatanga L, Rich T. E-learning and educational diversity. Nurse Educ Today. 2002 Jan;22(1):76-82; discussion 83-4. doi: 10.1054/nedt.2001.0740. PMID 11886234
- [Result] Hester L, Reed B, Bohannan W, Box M, Wells M, O'Neal B. Using an educational mobile application to teach students to take vital signs. Nurse Educ Today. 2021 Dec;107:105154. doi: 10.1016/j.nedt.2021.105154. Epub 2021 Sep 16. PMID 34583238
- [Result] Johnson N, List-Ivankovic J, Eboh WO, Ireland J, Adams D, Mowatt E, Martindale S. Research and evidence based practice: using a blended approach to teaching and learning in undergraduate nurse education. Nurse Educ Pract. 2010 Jan;10(1):43-7. doi: 10.1016/j.nepr.2009.03.012. Epub 2009 May 6. PMID 19423398
- [Result] Kenny A. Online learning: enhancing nurse education? J Adv Nurs. 2002 Apr;38(2):127-35. doi: 10.1046/j.1365-2648.2002.02156.x. PMID 11940125
- [Result] Kim JH, Park H. Effects of Smartphone-Based Mobile Learning in Nursing Education: A Systematic Review and Meta-analysis. Asian Nurs Res (Korean Soc Nurs Sci). 2019 Feb;13(1):20-29. doi: 10.1016/j.anr.2019.01.005. Epub 2019 Jan 16. PMID 30659927
- [Result] Lee NJ, Chae SM, Kim H, Lee JH, Min HJ, Park DE. Mobile-Based Video Learning Outcomes in Clinical Nursing Skill Education: A Randomized Controlled Trial. Comput Inform Nurs. 2016 Jan;34(1):8-16. doi: 10.1097/CIN.0000000000000183. PMID 26389858
- [Result] O'Connor S, Andrews T. Smartphones and mobile applications (apps) in clinical nursing education: A student perspective. Nurse Educ Today. 2018 Oct;69:172-178. doi: 10.1016/j.nedt.2018.07.013. Epub 2018 Aug 1. PMID 30096510
- [Result] Rose S. Medical Student Education in the Time of COVID-19. JAMA. 2020 Jun 2;323(21):2131-2132. doi: 10.1001/jama.2020.5227. No abstract available. PMID 32232420
- [Result] Shen WQ, Chen HL, Hu Y. The validity and reliability of the self-directed learning instrument (SDLI) in mainland Chinese nursing students. BMC Med Educ. 2014 May 27;14:108. doi: 10.1186/1472-6920-14-108. PMID 24885557
- [Result] Thiele JE. Learning patterns of online students. J Nurs Educ. 2003 Aug;42(8):364-6. doi: 10.3928/0148-4834-20030801-08. PMID 12938899
- [Result] Willemse JJ, Bozalek V. Exploration of the affordances of mobile devices in integrating theory and clinical practice in an undergraduate nursing programme. Curationis. 2015;38(2):e1-e10. doi: 10.4102/curationis.v38i2.1510. Epub 2015 Sep 28. PMID 26852423